CLINICAL TRIAL: NCT01832025
Title: Comparison of the Intraoperative, Postoperative Complications and Patient's Discomfort Involving External and Internal Maxillary Sinus Floor Elevation Techniques With Simultaneous Implant Placement: a Randomized Clinical Trial
Brief Title: Comparison of Incidence Between Two Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUSDM10665; 10665 (Other: Tufts University IRB)
Record Dates: First submitted 2013-04-08; First posted 2013-04-15 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Edentulous Posterior Maxilla
Keywords: intraoperative; postoperative; complications; discomfort; external; internal; maxillary; elevation; implant; reconstruction; bone; sinus
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internal (Active Comparator): internal maxillary sinus floor elevation technique with simultaneous implant placement
  Interventions: Procedure: internal maxillary sinus floor elevation technique
- External (Active Comparator): external maxillary sinus floor elevation technique with simultaneous implant placement
  Interventions: Procedure: external maxillary sinus floor elevation technique

INTERVENTIONS:
Procedure: internal maxillary sinus floor elevation technique — The internal lift procedure uses a drilling instrument (a drill that cuts through bone) to break through the bone for where the implant will later go. This creates an opening in the necessary area to allow more bone material to be added, which will move the sinus up and allow for the implant to be securely placed.
  Arms: Internal
Procedure: external maxillary sinus floor elevation technique — The external lift procedure involves cutting through the upper-most part of the gums to then cut through the bone to create an opening in the necessary area. The sinus will be manually lifted and the bone material will be added, which will allow for the implant to be securely placed.
  Arms: External

SUMMARY:
Sinus augmentation, also referred to as a sinus lift or a sinus graft, is an oral surgery procedure where bone is added to the upper jaw near the molars. The goal of the surgery is to add enough bone material onto the upper jaw to support the placement of a dental implant. The augmentation and the dental implant placement will be done at the same time to avoid the need for two surgeries. This is standard of care.

The purpose of this study is to compare any problems and patient comfort levels following surgery. Subjects will be randomly placed into one of two groups: the internal lift group or the external lift group. Both types of surgery are routinely done at our clinic. Usually the type of procedure (internal or external) is based on the dentist's preference. Investigators are doing this study to compare them to each other to see if one is more comfortable for the subject than the other or if they are equal. It is predicted that the two techniques may differ when it comes to complications during the procedure, patient discomfort following the procedure and patient complications in the weeks and months after the procedure. This last comparison has not yet been studied, and surgeons often choose the technique that they prefer from their own experiences. With this research study researchers hope to gain valuable information that will help surgeons' decisions in the future.

* Investigators hypothesize that external sinus augmentation with simultaneous implant placement (external technique) will have a higher rate of Schneiderian membrane perforation than the internal sinus augmentation with simultaneous implant placement (internal technique).
* Investigators hypothesize that the internal technique is associated with more discomfort for the subject compared with the external technique.
* Investigators hypothesize that the external technique will result in more severe pain/bleeding/swelling than the internal technique.
* Investigators hypothesize that the internal technique has a higher incidence of complications that occur between three weeks and three months postoperatively compared with the external technique.
* Investigators hypothesize that the external technique has a higher amount of analgesics taken postoperatively compared with the internal technique

DETAILED DESCRIPTION:
Experimental Design

The proposed study design is a single site, double armed, randomized clinical trial. Subjects will be those whose diagnosis requires restoring the lateral maxillary edentulous area by performing sinus augmentation together with implant placement.

Sample Size and Statistical Analysis Sample size A number of 46 subjects, 23 per each group, who meet study inclusion and exclusion criteria, will be treated for this study to allow for a dropout rate of up to 15%. Up to 60 subjects will be consented to reach the research goal of 46.

The sample size was determined using nQuery program (version 7.0) - for a power of 80% with 20 subjects/group, assuming the anticipated values for the Schneiderian membrane rate perforation as 55% (8) for the external procedure and 10% for the internal procedure (9), based on previously reported studies for each procedure.

Randomization Randomization will be performed in a 1:1 ratio using a balanced design based on a computer-generated randomization scheme. A printout of this scheme will be used by the co-investigator which will have the randomization for each subject that qualifies in the order of qualification. Randomization will occur the day of surgery.

Blinding Due to the nature of the procedures, this study will not be blinded.

Subject Characteristics Subjects will include patients whose diagnosis requires restoring the lateral maxillary edentulous area by performing sinus augmentation together with implant placement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* patients treatment planned for sinus lift augmentation and implant placement, with a height of the crestal alveolar bone measured in the middle of the edentulous space between four and six mm (calibrated measurements recorded on existing panoramic radiograph)
* the length of the edentulous span is one or two teeth
* non-smokers

Exclusion Criteria:

* patients who have had a previous sinus lift augmentation procedure
* pathology present within the sinus (sinusitis, polyps, neoplasia, mucoceles, etc.) or any deformity/radiation therapy to the sinus
* medically compromised patients contraindicated to dental surgery at TUSDM periodontal clinic including uncontrolled diabetes (HbA1c ≥7, lab results from within the past 6 months will be reviewed, patient without lab results from within the past 6 months will be excluded) and/or uncontrolled hypertension (more than stage II, ≥160/110)
* patients with medical condition that could potentially affect wound healing (e.g., self-reported Hepatitis B or C, self-reported HIV)
* patients with metabolic bone disease such as Paget's Disease or osteoporosis
* patients who are currently taking bisphosphonates or steroids
* patients who are currently pregnant according to self-report (standard of care in the TUSDM Periodontology clinic for such procedures)
* current smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Compare incidence of Schneiderian membrane perforation | 1-3 months after surgical procedure
  Compare the incidence of Schneiderian membrane perforation involving sinus augmentation interventions - external and internal technique with simultaneous implant placement.

SECONDARY OUTCOMES:
Compare discomfort | 1-3 months after surgical procedure
  Compare the subject's discomfort during both procedures using a validated survey form filled in by the subject at the end of the procedure.
Compare long term complications | 3 weeks to 3 months after surgical procedure
  Compare the long term complications that occur after both procedures, evaluated after three weeks and three months. This includes pain, bleeding, swelling or any other adverse events that the subject has experienced related to the procedures being observed.
Compare the amount of analgesic taken postoperatively | 1-3 months after surgical procedure
  Compare the amount of analgesic taken postoperatively evaluated using a subject's medication log.
Compare pain | 1 week after surgical procedure
  Compare the severity of pain between the two groups, one week after the procedures, using a validated survey.
Compare Bleeding | One week after surgical procedure
  Compare the severity of bleeding between the two groups, one week after the procedures, using a validated survey.
Compare Swelling | One week after surgical procedure
  Compare the severity of swelling between the two groups, one week after the procedures, using a validated survey.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Hur, DMD MS, Principal Investigator — TUSDM
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No